CLINICAL TRIAL: NCT06422182
Title: Ultrasound-Guided Erector Spinae Plane Block in Radical Cystectomy: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block in Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Tarek Ezzat Abd El Galil, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2112-301-058
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Erector Spinae Plane Block; Radical Cystectomy
MeSH Terms: interventions — Morphine; Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block group (Experimental): Patients received ultrasound guided bilateral single shot erector spinae pane block (ESPB) at Th10 level with 20 mL 0.25% bupivacaine after the end of surgery.
  Interventions: Drug: Bupivacain 25% (Erector Spinae Plane Block)
- Intravenous patient-controlled analgesia group (Active Comparator): Patients received Intravenous patient-controlled analgesia (IV-PCA) by morphine
  Interventions: Drug: Morphine (Intravenous patient-controlled analgesia)

INTERVENTIONS:
Drug: Bupivacain 25% (Erector Spinae Plane Block) — Patients received ultrasound guided bilateral single shot erector spinae pane block (ESPB) at Th10 level with 20 mL 0.25% bupivacaine after the end of surgery.
  Arms: Erector Spinae Plane Block group
Drug: Morphine (Intravenous patient-controlled analgesia) — Patients received intravenous patient-controlled analgesia (IV-PCA) by morphine
  Arms: Intravenous patient-controlled analgesia group

SUMMARY:
The aim of this research is to study and compare the efficacy and safety of bilateral single injection erector spinae plane block (ESPB) compared with intravenous patient-controlled analgesia (IV-PCA) in managing postoperative pain after radical cystectomy.

DETAILED DESCRIPTION:
Radical cystectomy (RC) is one of the most challenging surgical techniques in Urology. Acute postsurgical pain is frequently detrimental in a patient's recovery and quality of life.

Intravenous patient-controlled analgesia (IV-PCA) is one of the most commonly used strategies in clinical practice for controlling postoperative pain. It involves continuous administration of a programmed dose of analgesics, while also allowing patients to receive additional, need-based doses.

One such avenue is the erector spinae plane block (ESPB), a novel analgesic technique first described in 2016 by Forero et al. Although the mechanism of action of the ESPB is unknown, a proposed mechanism is via blockade of the dorsal and ventral rami of thoracic/lumbar spinal nerves. ESPB has been used as analgesia in rib fractures and other thoracic procedures as well as in abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient between 21 to 65 years.
* Both sexes.
* Body mass index (BMI): 20 - 40 kg/m2.
* American Society of Anesthesiologists (ASA) physical status II-III.
* Elective radical cystectomy.

Exclusion Criteria:

* Patient refusal.
* Psychiatric and cognitive disorders.
* Local infection at the site of injection.
* Allergy to study medications.
* Anatomic abnormalities.
* Inability to comprehend or participate in pain scoring system.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  Bolus dose of IV morphine (3mg) was provided as a rescue analgesia when the numeric rating scale (NRS) ≥ 4.

SECONDARY OUTCOMES:
The time of first rescue analgesia | 48 hours postoperatively
  Time from end of surgery to first dose of morphine administrated.
Degree of pain | 48 hours postoperatively
  Pain assessment will be done at rest and during coughing or movement by numeric rating scale (NRS) from 0 to 10 where 0 means no pain and 10 being worst pain) at PACU, 2, 4, 8, 12, 16 24, 36 and 48 postoperative.
Incidence of side effects | 48 hours postoperatively
  Side effects such as hypotension, bradycardia, respiratory depression (respiratory rate <10/minute), urinary retention and postoperative nausea and vomiting (PONV) will be recorded and managed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.